CLINICAL TRIAL: NCT06844578
Title: Assessment of Postural Control and Balance in the Older Adult
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Alejandro Caña Pino, Clinical Proffesor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 160225
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Older Adult; Balance Assessment; Older Adults, Balance; Postural Balance
Keywords: postural control; assessment; older adult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (G1) or control (No Intervention): This group will be composed of 20 participants who will not receive any spe
- Group 2 (G2) or active comparator (Active Comparator): will consist of 20 participants who will receive an intervention based exclusively on gerontogymnastics.
  This programme will include a series of exercises adapted to the needs of the older adult population, with emphasis on improving balance, muscle strength, flexibility and motor coordination.
  motor coordination.
  Interventions: Other: Active comparator Group
- Group 2 (G2) or experimental (Experimental): will consist of 20 participants who will receive a combined combined intervention. This will consist of a programme of gerontogymnastics, and a specific occupational therapy plan, in which exercises will be carried out, such as which will include exercises such as: Unipodal Stability, Gait Re-education, Muscle Strength, Stationary Gait.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — specific intervention programme in the experimental group, which will be carried out over a period of 6 weeks, with a total of 12 scheduled sessions of 45 minutes each. The programme will be aimed at improving various functional capacities, through specifically designed exercises, including:
  * Unipodal stability: Exercises focused on strengthening balance by maintaining a posture on one foot, which is key to preventing falls and improving postural stability.
  * Gait re-education: Activities aimed at correcting and adjusting gait technique, promoting an efficient and safe movement pattern.
  * Muscle strength: Exercises aimed at muscle strengthening, especially in the lower limbs, to increase endurance and stability during daily activities.
  * Stationary walking: Practices that simulate stationary walking, improving cardiovascular endurance and motor coordination.
  Arms: Group 2 (G2) or experimental
Other: Active comparator Group — which will be carried out over a period of 6 weeks, with a total of 12 scheduled sessions of 45 minutes each. Participants who will exclusively receive an intervention based on gerontogymnastics.
  This programme will include a series of exercises adapted to the needs of the older adult population, with an emphasis on improving balance, muscle strength, flexibility and motor coordination. These include:
  * Shoulder raises
  * Hip flexion
  * Knee flexion
  * Trunk rotations
  * Ankle dorsiflexion
  Arms: Group 2 (G2) or active comparator

SUMMARY:
A randomised clinical trial is proposed, using a probabilistic allocation design to ensure an equitable distribution of participants between the different intervention and control groups, minimising bias and increasing the internal validity of the results.

The trial foresees the voluntary participation of a total of 60 subjects, selected on the basis of previously established criteria and meeting specific characteristics criteria previously established and who meet the specific characteristics required for the study. The distribution of the participants in the clinical trial will be structured into three groups with characteristics and specific objectives, among which the following groups are highlighted:

* Group 1 (G1) or control: This group will be composed of 20 participants who will not receive any specific intervention related to gerontogymnastics or occupational therapy programmes designed from occupational therapy.
* Group 2 (G2) or experimental with gerontogymnastics: this group will be made up of 20 participants who will receive exclusively an intervention based on gerontogymnastics.

This programme will include a series of exercises adapted to the needs of the older adult population, with an emphasis on population, with emphasis on improving balance, muscle strength, flexibility and motor coordination.

Group 3 (G3) or experimental: will be composed of 20 participants who will receive a combined intervention. This will consist of a gerontogymnastics programme, mentioned above, merged with a specific occupational therapy plan, in which exercises such as:

* Unipodal stability
* Gait re-education
* Muscle strength
* Stationary gait

ELIGIBILITY:
Inclusion Criteria:

* Over 65 years old
* Residents Ntra. Sra. Del Rosario (Cáceres)
* Consent to participate
* Stable standing
* Tinetti <25

Exclusion Criteria:

* Does not meet inclusion criteria
* Medical contraindication to physical exercise
* Wheelchair mobility
* Severe cognitive impairment (>10 Minimental)
* VAS>4

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 6 weeks
  The MMSE is used to assess global cognitive function, identifying possible deficits in memory, language, orientation and attention on a scale from 0 to 30, where 30 indicates global cognitive function, and 0 may indicate severe cognitive impairment.
Visual Analogue Scale (VAS) | 6 weeks
  The VAS is a tool used to measure the level of pain intensity perceived by the patient. It allows participants to rate pain on a numerical scale from 0 to 10, with 0 being no pain and 10 being the maximum intensity.
Daniels Test | 6 weeks
  This test is intended to assess muscle function, specifically the gluteus maximus, quadriceps and hamstrings. It is used to determine the strength and endurance of these muscles in relation to postural stability and gait on a scale of 0 to 5, where 0 indicates no strength or inability to perform the movement and 5 indicates normal strength or optimal muscle function.
Timed Up and Go (TUG) | 6 weeks
  The TUG is an assessment method used to evaluate functional mobility and balance. It consists of measuring the time it takes for a subject to get up from a chair, walk three metres, turn around and sit down again.
Borg Scale | 6 weeks
  The Borg scale is used to measure the subjective perception of physical exertion during an activity. Participants rate their perception of fatigue as a function of exertion on a scale of 0 to 10.
Tinetti test | 6 weeks
  The Tinetti is a tool designed to assess the risk of falls in older adults. It examines postural stability and gait, allowing the identification of balance and mobility deficits that could compromise patient safety.
Functional Independence Measure (FIM) | 6 weeks
  The FIM is used to assess a patient's functional independence in various activities of daily living (ADLs), such as grooming, mobility and communication. It is a key tool for measuring functionality-related quality of life.
Joint position sense (JPS) | 6 weeks
  Assesses lumbar proprioceptive repositioning error using the IPhone inclinometer. Degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Enfermería y Terapia Ocupacional, Cáceres, Cáceres, Spain